CLINICAL TRIAL: NCT00080236
Title: Safety, Tolerability and Efficacy Study of a Caspase Inhibitor, IDN-6556, in Patients Undergoing Orthotopic Liver Transplantation (OLT)
Brief Title: Safety and Efficacy Study of a Caspase Inhibitor in Patients Undergoing Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Collaborators: Idun Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-000006556-PRO-0006
Record Dates: First submitted 2004-03-24; First posted 2004-03-26 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Liver Transplantation; Hepatitis; Cholestasis; Carcinoma, Hepatocellular
Keywords: Liver Transplantation
MeSH Terms: conditions — Hepatitis; Cholestasis; Carcinoma, Hepatocellular | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Donor organ placebo and Recipient placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Donor organ: IDN-6556 (15μg/ml), Recipient: Placebo (Active Comparator)
  Interventions: Drug: IDN-6556; Drug: Placebo
- Donor organ: IDN-6556 (5 μg/ml), Recipient: IDN-6556 0.5 mg/kg (Active Comparator)
  Interventions: Drug: IDN-6556
- Donor organ: IDN-6556(15 μg/ml), Recipient: IDN-6556 0.5 mg/kg (Active Comparator)
  Interventions: Drug: IDN-6556

INTERVENTIONS:
Drug: IDN-6556
  Arms: Donor organ: IDN-6556 (15μg/ml), Recipient: Placebo; Donor organ: IDN-6556 (5 μg/ml), Recipient: IDN-6556 0.5 mg/kg; Donor organ: IDN-6556(15 μg/ml), Recipient: IDN-6556 0.5 mg/kg
Drug: Placebo
  Arms: Donor organ placebo and Recipient placebo; Donor organ: IDN-6556 (15μg/ml), Recipient: Placebo

SUMMARY:
The purpose of the study is to test the safety and effectiveness of IDN-6556 in preventing liver damage that normally occurs when livers are transported before being transplanted and in the immediate post-transplant period.

DETAILED DESCRIPTION:
The occurrence of apoptosis in liver ischemia/reperfusion injury has been well characterized in animal models. In this context apoptosis has specifically been observed in sinusoidal endothelial cells and hepatocytes, and this has also been associated with an increase in activated caspase-3 in liver tissue extracts. The use of caspase inhibitors to prevent apoptosis during liver storage and transplantation may reduce ischemia/reperfusion injury and hence improve graft function after transplantation. Suppression of apoptosis by caspase inhibitors may also allow for longer ischemic times allowing organs to be transported greater distances. In addition, suppression of apoptosis may lower the risk involved in using suboptimal donor organs.

ELIGIBILITY:
Inclusion Criteria:

* Minimum adult age

Exclusion Criteria:

* Fulminant hepatic failure (UNOS Status I patients)
* Previous liver transplantation
* Patients undergoing split liver grafts
* Extrahepatic malignancy
* If female, pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2003-11; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Peak absolute change in alanine aminotransferase (ALT) values measured from baseline to up to 3 days post-transplantation
Peak absolute change in aspartate transaminase (AST) values measured from baseline to up to 3 days post-transplantation

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Mayo Clinic Scottsdale, Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Indiana University Medical Center, Indianapolis, Indiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Baylor Regional Transplant Institute, Baylor University Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Germany (3):
  - Oberarzt der Klinik für Allgemein-, Viszeral- und Transplantationschirurgie Charité-Virchow, Berlin
  - Klinik für Viszeral- und Transplantationschirurgie Medizinische Hochschule Hannover, Hanover
  - Abteilung für Transplantationschirurgie Johannes Gutenberg-Universität Mainz, Mainz